CLINICAL TRIAL: NCT07079462
Title: A Prospective Randomized Controlled Study Comparing 68Ga-FAPI PET-Guided Abdominal Radiotherapy Combined With Second-Line Standard Therapy and Cadonilimab Versus Second-Line Standard Therapy in Colorectal Cancer With Peritoneal Metastasis
Brief Title: Comparing 68Ga-FAPI PET-Guided Abdominal Radiotherapy Combined With Second-Line Standard Therapy and Cadonilimab Versus Second-Line Standard Therapy in Colorectal Cancer With Peritoneal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Dr, MD, PHD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TORCH-PM
Record Dates: First submitted 2025-07-12; First posted 2025-07-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Peritoneal (Metastatic) Cancer; FAPI PET
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy+Immunotherapy+Standard second-line systemic therapy (Experimental): Radiotherapy: The prescribed dose is 20-25Gy in 5 daily fractions to all or part of the target lesions.
  Immunotherapy: One week after the completion of radiotherapy, standard chemotherapy with cadonilimab, 6 mg/kg, is administered every two weeks.
  Standard second-line systemic therapy: Standard second-line systemic therapy: (XELOX/FOLFOX or XELIRI/FOLFIRI ± bevacizumab/cetuximab)
  Interventions: Combination Product: Radiotherapy followed by immunotherapy and chemotherapy
- Standard second-line systemic therapy (Active Comparator): Standard second-line systemic therapy: (XELOX/FOLFOX or XELIRI/FOLFIRI ± bevacizumab/cetuximab)
  Interventions: Drug: Chemotherapy (control)

INTERVENTIONS:
Combination Product: Radiotherapy followed by immunotherapy and chemotherapy — Radiotherapy: The prescribed dose is 20-25Gy in 5 daily fractions to all or part of the target lesions.
  Immunotherapy: One week after the completion of radiotherapy, standard chemotherapy with cadonilimab, 6 mg/kg, is administered every two weeks.
  Standard second-line systemic therapy: Standard second-line systemic therapy: (XELOX/FOLFOX or XELIRI/FOLFIRI ± bevacizumab/cetuximab)
  Arms: Radiotherapy+Immunotherapy+Standard second-line systemic therapy
Drug: Chemotherapy (control) — Standard second-line treatment regimen: (XELOX/FOLFOX or XELIRI/FOLFIRI ± bevacizumab/ cetuximab)
  Arms: Standard second-line systemic therapy

SUMMARY:
Main objective:

1. To compare the objective response rate (ORR) of 68Ga-FAPI PET-guided abdominal region radiotherapy combined with second-line standard treatment versus cabozantinib and second-line standard treatment in the treatment of peritoneal metastasis of colorectal cancer.

Secondary objectives:

1. To compare the disease control rate (DCR), duration of continuous remission (DoR), progression-free survival (PFS), and overall survival (OS) of 68Ga-FAPI PET-guided abdominal region radiotherapy combined with second-line standard treatment versus cabozantinib and second-line standard treatment in the treatment of peritoneal metastasis of colorectal cancer.
2. To evaluate the safety and tolerability of 68Ga-FAPI PET-guided abdominal region radiotherapy combined with second-line standard treatment versus cabozantinib.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of 18 years or older. 2. Peritoneal metastasis of colorectal cancer confirmed by histological or cytological examination (International Union Against Cancer 8th edition of colorectal cancer staging).

  3. Progression after receiving standard first-line treatment before enrollment; but excluding any type of immunotherapy.

  4. Eastern Cooperative Oncology Group (ECOG) score of 0-1, with an expected survival time of more than 6 months.

  5. ECOG score of 0-1. 6. Expected survival time of ≥ 24 weeks. 7. Laboratory tests for bone marrow, liver and kidney organ functions and coagulation function within 7 days before the first administration were in compliance with the study requirements (no blood transfusion, blood products, use of granulocyte colony-stimulating factor or other hematopoietic stimulating factors for correction within 7 days before the laboratory tests).

  8. Women with reproductive capacity must have a negative blood pregnancy test result within 7 days before the first administration. Male or female patients with reproductive capacity voluntarily use effective contraceptive methods during the study period and within 6 months after the last study medication, such as double barrier contraceptive methods, condoms, oral or injectable contraceptive drugs, intrauterine devices, abstinence, etc. All female patients will be considered to have reproductive capacity, unless the female patient has naturally menopause, artificial menopause or sterilization (uterus removal, bilateral ovary removal).

  9. Voluntary enrollment and signing of informed consent form, following the trial treatment plan and visit schedule.

Exclusion Criteria:

* 1. Absolute neutrophil count (ANC) < 1.5 × 109/L, or platelet count < 100 × 109/L (for patients with liver metastasis, platelet count < 80 × 109/L), or hemoglobin < 9 g/dL; blood transfusion within 2 weeks prior to enrollment is not allowed to meet the inclusion criteria.

  2. Serum total bilirubin > 1.5 times the upper limit of normal (ULN); for patients with liver metastasis, > 2.5 times ULN.

  3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 times ULN, or for patients with liver metastasis, ALT and/or AST > 5 times ULN.

  4. Serum creatinine > 1.5 times ULN, or creatinine clearance rate < 50 ml/min (calculated according to the Cockcroft-Gault formula).

  5. Partial thromboplastin time (APTT) or prothrombin time (PT) > 1.5 times ULN (based on the normal values of the clinical trial center).

  6. The researcher determines clinically significant severe electrolyte abnormalities.

  7. Urine protein test of 2+ or above, or 24-hour urine protein quantification ≥ 1.0 g/24h.

  8. Hypertension that is not well controlled by medication, defined as: systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg.

  9. The patient currently has active peptic ulcer, ulcerative colitis, or other digestive tract diseases or active bleeding from an unresected tumor, or the researcher determines that it may cause gastrointestinal bleeding or perforation; or if there was a previous gastrointestinal perforation or gastrointestinal fistula, and the patient has not recovered after surgical treatment.

  10. Within 6 months before enrollment, there is a history of arterial thrombosis or deep vein thrombosis, or within 2 months before enrollment, there is evidence or history of bleeding tendency or history of bleeding, regardless of severity.

  11. Within 12 months before enrollment, a stroke event or transient ischemic attack occurred.

  12. Within 6 months before enrollment, heart disease including congestive heart failure, acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass surgery; or NYHA class 2 or above heart dysfunction patients; left ventricular ejection fraction (LVEF) < 50%.

  13. Uncontrolled malignant pleural effusion, ascites or pericardial effusion (defined as not being effectively controlled by diuretics or puncture as determined by the researcher).

  14. Any patient who has received any anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibody (or any other antibody acting on the T cell co-stimulation or checkpoint pathways) before enrollment.

  15. Within 4 weeks before enrollment, received any form of radiotherapy. 16. At the screening stage, there is a clinically detectable second primary malignant tumor, or other malignant tumors occurred in the past 5 years, excluding fully treated non-melanoma skin cancer, cervical carcinoma in situ and superficial bladder tumor [non-invasive tumors, carcinoma in situ and T1 (tumor invasion of the lamina propria)], if present.

  17. Known clinical significance of liver disease history, including but not limited to known hepatitis B virus (HBV) infection and positive HBV DNA (≥ 1 × 104/ml); known hepatitis C virus (HCV) infection and positive HCV RNA (≥ 1 × 103/ml), or liver cirrhosis, etc.

  18. Pregnant or lactating women or women with a possibility of pregnancy who have a positive pregnancy test before the first medication; or female participants who are unwilling to implement strict contraception during the study.

The researcher considers that the subject has any clinical or laboratory abnormalities or non-compliance issues that make them unsuitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
ORR | From enrollment to the end of two treatment courses (each cycle is 14 days)
  After two treatment courses, the tumor shrinkage was evaluated according to the RECIST v1.1 standard. The therapeutic response was classified as PR/CR. Chemotherapy combined with immunotherapy (at the patient's expense) was continued, and it was denied to be stopped.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No